CLINICAL TRIAL: NCT03822741
Title: Gene Profiling and Individualized Treatment of Neonatal Seizure in China
Brief Title: Etiology and Treatment of Neonatal Seizure
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: CHFudanU_NNICU10
Record Dates: First submitted 2018-12-02; First posted 2019-01-30 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Seizures; Seizure Disorder; Seizure Newborn; Seizure Generalized
Keywords: seizure
MeSH Terms: conditions — Seizures; Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biological samples contain 2ml of blood, which is used to extract DNA from the blood for gene sequencing.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Genetic diagnosis for neonates suffering from epilepsy has important implications for treatment, prognosis, and development of precision medicine strategies. Investigator performed exome sequencing (ES) or targeted sequencing on neonates with seizure onset within the first month of life. Investigator subgrouped our patients based on the onset age of seizure into neonatal and before 1 year (1-12 months), to compare the clinical and genetic features and treatment strategies.

DETAILED DESCRIPTION:
Seizure is one of the most common neurological conditions in neonates, and has substantial impact on patients'quality of life and social integration. Epileptic encephalopathy is characterized by refractory seizures, cognitive dysfunction, and poor prognosis. Despite the recent progress in technology, molecular diagnosis of neonates suffering from possible epileptic seizures can be challenging, due to genetic and phenotypic heterogeneities. A large number of specific pathogenic variations have been related to various forms of epilepsies. Next-generation sequencing (NGS) has significantly improved the molecular diagnosis for rare diseases. NGS focusing on genes known to be associated with human diseases is a practical approach as a first-tier assessment for patients with heterogeneous genetic background. In addition, currently medical therapy for seizure is not based on the etiology, but the clinical manifestations, and the main purpose is not to rescue the underlying diseases process, but just to reduce the likelihood of seizures occurrence. In this study, Investigator performed NGS on neonates with seizure onset before 1 year of age, to detect and quantify genetic variants, and assess existing therapeutic effects. Our findings will have important implications for the development of precision medicine strategies.

ELIGIBILITY:
Inclusion Criteria:

* severe seizures in neonates or generalized epilepsy or intractable epilepsy in infancy with generalized tonic-clonic seizures,
* seizures onset before 1 year of age,
* epileptic syndromes/epileptic-encephalopathies with unknown etiology.

Exclusion Criteria:

* Patients were excluded if they had traumas, central nervous system infections, hypoxic-ischemic encephalopathy, vascular events, systemic infections, and diagnosed metabolic disorders, and pathogenic copy-number variants were identified using array-based comparative genomic hybridization (CGH).

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The subjects were treated in the Department of Neonatology of Children Hospital of Fudan University. All samples in this study were collected with appropriate informed consent and approval of the ethics committee of Children's Hospital, Fudan University. The methods used in this study were carried out in accordance with the approved guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-08-08 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Mutation rate of common seizure genes | From the oneset of seizure to the genetic sequencing finish, the process may last up to 3 months.
  We'll get the genetic profiles of all neonates who had seizures during this period. The mutation rate of common variant gene was calculated by gene spectrum.
Rate of seizure free | From the onset of seizure to 6 months after the onset of seizure
  After the onset of seizure, through clinical management and individualized intervention, we expect to observe the number and proportion of effective seizure treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhao Zhou, Doctor, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] EpiPM Consortium. A roadmap for precision medicine in the epilepsies. Lancet Neurol. 2015 Dec;14(12):1219-28. doi: 10.1016/S1474-4422(15)00199-4. Epub 2015 Sep 20. PMID 26416172
- [Background] Lemke JR, Riesch E, Scheurenbrand T, Schubach M, Wilhelm C, Steiner I, Hansen J, Courage C, Gallati S, Burki S, Strozzi S, Simonetti BG, Grunt S, Steinlin M, Alber M, Wolff M, Klopstock T, Prott EC, Lorenz R, Spaich C, Rona S, Lakshminarasimhan M, Kroll J, Dorn T, Kramer G, Synofzik M, Becker F, Weber YG, Lerche H, Bohm D, Biskup S. Targeted next generation sequencing as a diagnostic tool in epileptic disorders. Epilepsia. 2012 Aug;53(8):1387-98. doi: 10.1111/j.1528-1167.2012.03516.x. Epub 2012 May 21. PMID 22612257
- [Background] Moller RS, Larsen LH, Johannesen KM, Talvik I, Talvik T, Vaher U, Miranda MJ, Farooq M, Nielsen JE, Svendsen LL, Kjelgaard DB, Linnet KM, Hao Q, Uldall P, Frangu M, Tommerup N, Baig SM, Abdullah U, Born AP, Gellert P, Nikanorova M, Olofsson K, Jepsen B, Marjanovic D, Al-Zehhawi LI, Penalva SJ, Krag-Olsen B, Brusgaard K, Hjalgrim H, Rubboli G, Pal DK, Dahl HA. Gene Panel Testing in Epileptic Encephalopathies and Familial Epilepsies. Mol Syndromol. 2016 Sep;7(4):210-219. doi: 10.1159/000448369. Epub 2016 Aug 20. PMID 27781031
- [Background] Striano P, Zara F. Epilepsy: Common and rare epilepsies share genetic determinants. Nat Rev Neurol. 2017 Apr;13(4):200-201. doi: 10.1038/nrneurol.2017.30. Epub 2017 Mar 10. No abstract available. PMID 28281535
- [Background] Striano P, Vari MS, Mazzocchetti C, Verrotti A, Zara F. Management of genetic epilepsies: From empirical treatment to precision medicine. Pharmacol Res. 2016 May;107:426-429. doi: 10.1016/j.phrs.2016.04.006. Epub 2016 Apr 11. PMID 27080588
- [Background] Wang K, Li M, Hakonarson H. ANNOVAR: functional annotation of genetic variants from high-throughput sequencing data. Nucleic Acids Res. 2010 Sep;38(16):e164. doi: 10.1093/nar/gkq603. Epub 2010 Jul 3. PMID 20601685
- [Background] Myers CT, Mefford HC. Advancing epilepsy genetics in the genomic era. Genome Med. 2015 Aug 25;7(1):91. doi: 10.1186/s13073-015-0214-7. PMID 26302787